CLINICAL TRIAL: NCT04901429
Title: Truncal Vagotomy in Patients Undergoing Revisional Sleeve Gastrectomy to Gastric Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 021-171
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Vagotomy, Truncal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Truncal Vagotomy (Experimental): Truncal vagotomy will be performed during other routine procedure.
  Interventions: Procedure: Truncal vagotomy
- No Truncal Vagotomy (No Intervention): No truncal vagotomy will be performed during other routine procedure.

INTERVENTIONS:
Procedure: Truncal vagotomy — Truncal vagotomy will be performed in 50% of patients during other routine procedure.
  Arms: Truncal Vagotomy

SUMMARY:
The purpose of this study is to investigate the efficacy of performing a truncal vagotomy along with a sleeve to bypass revision surgery in reducing the severity and/or incidence of gastroesophageal reflux disease (GERD) post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participating subjects will need to be >18yrs of age and eligible for sleeve to bypass revision bariatric surgery.
* Undergoing sleeve to bypass revision bariatric surgery.

Exclusion Criteria:

* Patients who are under the age of 18.
* Not eligible for sleeve to bypass revision bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
GERD-HRQL scores | approximately 6 months post operation
  GERD-HRQL scores
Esophageal pH monitoring | approximately 6 months post operation
  Esophageal pH monitoring
Reflux symptom index questionnaire | approximately 6 months post operation
  Reflux symptom index questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided